

# TRIAL STATISTICAL ANALYSIS PLAN

c26461609-01

| BI Trial No.: | 1405-0001 |
|---|---|
| Title: | Safety, tolerability, pharmacokinetics, and pharmacodynamics of single rising oral doses of BI 1323495 in healthy male subjects (single-blind, partially randomised, placebo-controlled parallel group design) |
| | Including Protocol Amendment 1 and 2 [c21116620-03] |
| Investigational Product: | BI 1323495 |
| Responsible trial statisticians: | |
| | Phone:<br>Fax: |
| | Phone:<br>Fax: |
| Date of statistical analysis plan: | 10 JAN 2019 SIGNED |
| Version: | Final |

**Proprietary confidential information** 

© 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1405-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### TABLE OF CONTENTS 1.

| TITLE | PAGE | 1 |
|------------|------------------------------------------------|----|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | OF TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 8 |
| 5. | ENDPOINTS | 9 |
| 5.1 | PRIMARY ENDPOINTS | 9 |
| 5.2 | SECONDARY ENDPOINTS | |
| 5.2.1 | Key secondary endpoints | 9 |
| 5.2.2 | Secondary endpoints | |
| 6. | GENERAL ANALYSIS DEFINITIONS | 12 |
| 6.1 | TREATMENTS | |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS | 13 |
| 6.3 | SUBJECT SETS ANALYSED | 15 |
| 6.5 | POOLING OF CENTRES | 16 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | 16 |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | PLANNED ANALYSIS | 20 |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 22 |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | 22 |
| 7.3 | TREATMENT COMPLIANCE | 22 |
| 7.4 | PRIMARY ENDPOINTS | 22 |
| 7.5 | SECONDARY ENDPOINTS | 23 |
| 7.5.1 | Key secondary endpoints | 23 |
| 7.5.2 | Secondary endpoints | 23 |
| 7.7 | EXTENT OF EXPOSURE | 26 |
| <b>7.8</b> | SAFETY ANALYSIS | 26 |
| 7.8.1 | Adverse events | 26 |
| 7.8.2 | Laboratory data | 28 |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG | |
| 7.8.5 | Others | 30 |
| 8. | REFERENCES | 31 |

# **Boehringer Ingelheim**

| TSAP for | BI | Trial | No: | 1405-0001 |
|----------|----|-------|-----|-----------|
|----------|----|-------|-----|-----------|


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

10. HISTORY TABLE......36

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1405-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 | Labels for treatments for use in the CTR | 12 |
|--------------|----------------------------------------------|----|
| Table 6.2: 1 | Important protocol deviations | 14 |
| Table 6.3: 1 | Analysis sets for endpoints/data description | 16 |
| Table 10: 1 | History table | 36 |

TSAP for BI Trial No: 1405-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

| Term | Definition / description |
|---|---|
| ADS | Analysis Dataset |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ALT | Alanine Aminotransferase |
| ANCOVA | Analysis of Covariance |
| AST | Aspartate Aminotransferase |
| $AUC_{0\text{-}\infty}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity |
| BI | Boehringer Ingelheim |
| BMI | Body mass index |
| CI | Confidence Interval |
| $C_{max}$ | Maximum measured concentration of the analyte in plasma |
| CRF | Case Report Form |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic Coefficient of Variation |
| DB | Dose Proportionality, Between-Subject Design |
| DBLM | Database Lock Meeting |
| DILI | Drug induced liver injury |
| ECG | Electrocardiogram |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials |
| gCV | Geometric Coefficient of Variation |
| gMean | Geometric Mean |
| ICH | International Conference On Harmonisation |
| ISF | Investigators Site File |
| iPD | Important Protocol Deviation |
| LLT | Lower Level Term |

Boehringer Ingelheim
TSAP for BI Trial No: 1405-0001
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|---|---|
| Max | Maximum |
| MedDRA | Medical Dictionary For Regulatory Activities |
| Min | Minimum |
| N | Number non-missing observations |
| P10 | 10 <sup>th</sup> percentile |
| P90 | 90 <sup>th</sup> percentile |
| PD | Pharmacodynamic(s) |
| PK | Pharmacokinetic(s) |
| PKS | PK parameter analysis set |
| PT | Preferred Term |
| Q1 | 1 <sup>st</sup> quartile |
| Q3 | 3 <sup>rd</sup> quartile |
| QD | Quaque die, once daily |
| RAGe | Report Appendix Generator system |
| REP | Residual Effect Period |
| RPM | Report Planning Meeting |
| $\mathrm{SAS}^{\circledR}$ | Statistical Analysis System |
| SD | Standard Deviation |
| SOC | System Organ Class |
| t <sub>max</sub> | Time from dosing to maximum measured concentration of the analyte in plasma |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper Limit of Normal |
| WHO-DD | World Health Organization Drug Dictionary |
| XPKISTAT | Library of SAS® Macros for PK analysis |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 3. INTRODUCTION

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This trial statistical analysis plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data will be stored in a trial database within the RAVE EDC system.

Pharmacokinetic (PK) parameters will be calculated using

The statistical analyses will be performed within the validated working environment CARE, including SAS® (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SASTM-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses as planned in the CTP will be performed and are described in more detail in this TSAP. The following changes compared to the protocol will be made:

# 5. ENDPOINTS

### 5.1 PRIMARY ENDPOINTS

### **Section 5.2.1 of the CTP:**

Primary endpoint to assess safety and tolerability of BI 1323495 is the number [N (%)] of subjects with drug-related adverse events.

#### 5.2 SECONDARY ENDPOINTS

# 5.2.1 Key secondary endpoints

This section is not applicable as no key secondary endpoints have been defined in the CTP.

# 5.2.2 Secondary endpoints

### Section 5.5.1.1 of the CTP:

- $AUC_{0-\infty}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
- $C_{max}$  (maximum measured concentration of the analyte in plasma)

TSAP for BI Trial No: 1405-0001 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1405-0001 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

It is planned that in total 64 healthy male subjects will participate in this study, according to 8 sequential groups comprising 8 subjects per group. Within each dose group, 6 subjects will receive the active drug and 2 will receive placebo.

For details of dosage and formulation see Table 6.1:1 below.

Table 6.1: 1 Labels for treatments for use in the CTR

| Dose<br>group | Treatment | | | Short label |
|---|---|---|---|---|
| 1-8 | P* | Placebo, tablet, qd | | Placebo |
| 1 | A | BI 1323495, | tablet, po, qd | BI |
| 2 | В | BI 1323495, | tablet, po, qd | BI |
| 3 | C | BI 1323495, | tablet, po, qd | BI |
| 4 | D | BI 1323495, | tablet, po, qd | BI |
| 5 | E | BI 1323495, | tablet, po, qd | BI |
| 6 | F | BI 1323495, | tablet, po, qd | BI |
| 7 | G | BI 1323495, | tablet, po, qd | BI |
| 8 | Н | BI 1323495, | tablet, po, qd | BI |

<sup>\*:</sup> The placebo group in the safety evaluation will consist of all placebo treated subjects, regardless of the dose group in which they were treated.

The following separate study phases will be defined for the analyses of AEs:

- Screening (ranging from 0:00h (midnight) on day of informed consent until administration time of study drug (BI or Placebo))
- On treatment
  - o **BI/Placebo treatment** (separately for each treatment, ranging from the time of administration of BI / Placebo until 0:00h (midnight) on the day after trial completion date)

Please note that all AEs reported between start of trial drug administration and the last perprotocol contact will be considered on treatment (i.e. no follow-up period is considered in this trial).

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Two types of AE displays will be provided in the report:

**A)** Section 15.3 and Appendix 16.1.13.1.8 (for ClinicalTrials.gov and EudraCT) of the CTR displays:

In these displays, the on-treatment phase will be analysed (labelled with the name of the study treatment (short label)). Screening will not be included in this analysis. The following totals will be provided in addition:

- a total over all BI treated phases ("BI Total")
- a total over all on treatment phases included in this analysis ("**Total on treatment**") (Section 15.3 only)
- **B)** Section 15.4 and Appendix 16.1.13.1.8 (except for ClinicalTrials.gov and EudraCT) of the CTR displays:
  - Screening
  - On treatment (labelled with the name of the study treatment (short label))

In Section 16.1.13.1.8 AE tables, the following totals will be provided in addition:

- a total over all BI treated phases ("BI Total")
- a total over all study phases ("**Total**")

Tables of vital signs and laboratory values will present results by the above mentioned on treatment phase.

For detailed information on the handling of the treatments refer to Technical TSAP ADS (analysis data set) plan and Data Reviewers guide.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Data discrepancies and deviations from the CTP will be identified for all treated subjects.

Consistency check listings (for identification of deviations of time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the Report Planning Meeting and database lock meeting (RPM/DBLM). At this meeting, all manual deviations identified at the sites by the CRAs and deviations too complex to program will be reviewed by the trial team to decide which are considered important. For definition of important protocol deviations (iPD), and for the process of identification of these, refer to the Boehringer Ingelheim (BI) SOP "Identify and Manage Important Protocol Deviations (iPD)" (2).

If any iPDs are identified, they are to be summarised into categories and will be captured in the RPM/DBLM minutes via an accompanying Excel spreadsheet (3). The following table contains the categories which are considered to be iPDs in this trial. If the data show other iPDs, this table will be supplemented accordingly by the time of the RPM/DBLM at the latest.

Important protocol deviations will be summarised and listed.

Table 6.2: 1 Important protocol deviations

| Cate | gory/Code | Description |
|---|---|---|
| A | | Entrance criteria not met |
| | A1 | Inclusion criteria violated |
| | A2 | Exclusion criteria violated |
| В | | Informed consent |
| | B1 | Informed consent not available |
| | B2 | Informed consent too late |
| C | | Trial medication and randomisation |
| | C1 | Incorrect trial medication taken |
| | C2 | Randomisation not followed |
| | C3 | Non-compliance |
| | C4 | Incorrect intake of trial medication |
| D | | Concomitant medication |
| | D1 | Concomitant medication with the potential to affect the assessment of the trial medication |
| E | | Missing data * |
| | E1 | None |
| F | | Incorrect timing <sup>1</sup> |
| | F1 | Certain deviations from time schedule used to measure secondary data |
| G | | Other trial specific important deviations |
| | G1 | Incorrect intake of meal before administration of treatment |
| | G2 | Protocol deviations affecting safety and rights |

Time deviations will only be flagged as iPD, when leading to exclusion of the entire subject from an analysis set

<sup>\*</sup> Missing visits, evaluations, and tests will be considered missing data, not protocol deviations

### 6.3 SUBJECT SETS ANALYSED

• Treated set (TS):

This subject set includes all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment. This is the full analysis set population in the sense of ICH-E9 (1). It is used for demographics, baseline characteristics, and safety analyses, as well as for the description of biomarkers.

• PK parameter analysis set (PKS):

The PK parameter analysis set (PKS) includes all subjects from the TS receiving BI 1323495 who provide at least one secondary PK parameter that was not excluded according to the description below.

It is used for assessment of dose proportionality.

**Section 7.3.2 of the CTP:** Plasma concentration data and parameters of a subject will be included in the statistical PK analyses if they are not flagged for exclusion due to a protocol deviation relevant to the evaluation of PK (to be decided no later than in the RPM) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the CTR.

Relevant protocol deviations may be:

- Incorrect trial medication taken, i.e. the subject received at least one dose of trial medication the subject was not assigned to
- Incorrect dose of trial medication taken
- *Use of restricted medications*

Plasma concentrations and/or parameters of a subject will be considered as non-evaluable, if for example:

- The subject experienced emesis that occurred at or before two times median  $t_{max}$  of the respective treatment (median  $t_{max}$  is to be determined excluding the subjects experiencing emesis),
- Missing samples/concentration data at important phases of PK disposition curve.

The descriptive analysis of PK concentrations will be based on the ADS ADPC as described at the beginning of Section 7.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.3: 1 Analysis sets for endpoints/data description

| Endpoint/data description | TS | PKS |
|--------------------------------------|----|-----|
| Primary and further safety endpoints | X | |
| Description of biomarkers | X | |
| Secondary PK endpoints | | X |
| Demographic/baseline data | X | |
| Important protocol deviations | X | |
| Disposition | X | |

#### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Handling of missing data and outliers will be performed as described in the CTP, Section 7.4.

The only exceptions where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards (see 001-MCG-156\_RD-01 (4)).

Missing data and outliers of PK data are handled according to BI standards (see 001-MCS-36-472\_RD-01) (5).

# 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

The baseline value is defined as the last measurement before administration of BI 1323495 or Placebo.

**Section 6.1 of the CTP:** Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening and end of trial examination are given in the CTP Flow Chart.

Study measurements and assessments scheduled to occur 'before' trial medication administration on Day 1 are to be performed and completed within a 3 h-period prior to the trial drug administration (including blank values for PK and biomarkers).

Adherence to time windows will be checked via the consistency check listings at the RPM/DBLM.

Boehringer Ingelheim
TSAP for BI Trial No: 1405-0001
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| - | | | | | |
|---|---|----------|---|--------------|---|
| _ | | | | | _ |
| | | _ | | | |
| | | _ | | | |
| | | | | <del> </del> | |
| | | _ | _ | | |
| | | _ | | | |
| | | _ | | | |
| | | _ | _ | | |
| | | _ | | | |
| | | _ | | | |
| | | <u> </u> | | | |
| I | · | | | | |

TSAP for BI Trial No: 1405-0001 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 7. PLANNED ANALYSIS

The placebo group in the safety evaluation will consist of all placebo treated subjects, regardless of the dose group in which they were treated.

Safety analysis (refer to Section 7.8) will be performed by and will be presented in Sections 15.1 to 15.4 of the CTR and in Appendix 16.2 and 16.1.13.1.

Descriptive data analysis of PD parameters will be performed by and will be presented in Sections 15.7 of the CTR.

Inferential statistical analyses of PK and PD endpoints (refer to Section 7.5.2) will also be performed by and will be presented in Section 15.5, and 15.7 of the CTR and in Appendices 16.1.13.3 and 16.1.13.6.

Descriptive data analysis of PK parameters and concentrations will be performed by the department Translational Medicine and Clin. Pharmacology at BI and will be presented in Section 15.6 and 15.7 of the CTR.

The format of the listings and tables will follow the standards defined in the BI corporate guideline "Reporting of Clinical Trials and Project Summaries" [001-MCG-159] (6) with the exception of those generated for PK-calculations.

The individual values of all subjects will be listed, sorted by treatment group, subject number, and visit.

The listings will be included in Appendix 16.2 of the CTR.

For end-of-text tables, the set of summary statistics for non-PK parameters is:

N number non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For analyte concentrations, the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For PK parameters, the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

P10 10th percentile
Q1 1st quartile
Q3 3rd quartile
P90 90th percentile

The data format for descriptive statistics of concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category, as well as the percentage (%) for each treatment group. Percentages will be rounded to one decimal place and will be based on all subjects in the respective subject set whether they have non-missing values or not. The category 'missing' will be displayed only if there are actually missing values.

Units of variables should be given in the titles or column/row descriptors in square brackets (e.g. [mg]).

# Exclusion of PK parameters

The ADS ADPP (PK parameters) contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS will include parameters if they are not flagged for exclusion, that is APEXC is equal to "Included".

### Exclusion of PK concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to 'ALL CALC', the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to 'DESC STATS', the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition 'TIME VIOLATION' or 'TIME DEVIATION', the value can be used for further analyses based on actual times. If ACEXCO is set to 'HALF LIFE', the value will be excluded from half-life calculation (and, as a consequence, any calculation that relies on  $\lambda_z$ ) only; the value is included for all other analyses.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Further details are given in 001-MCS-36-472\_RD-01 "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (5) and 001-MCS-36-472\_RD-03 "Description of Analytical Transfer Files and PK/PD Data Files" (7).

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report, based on the TS.

The data will be summarised by treatment group and in total.

### 7.2 CONCOMITANT DISEASES AND MEDICATION

Frequency tables are planned for this section of the report, based on the TS.

Concomitant diseases will be coded using the latest version of the coding system of the Medical Dictionary for Drug Regulatory Activities (MedDRA). Medications will be coded using the latest version of the World Health Organization Drug Dictionary (WHO-DD). The coding version number will be displayed as a footnote in the respective output.

The diagnoses and medications will be listed. Subjects without any concomitant diagnoses or concomitant therapies should be marked with a "No" in the respective column.

The relevance of the concomitant therapies to the evaluation of PK will be decided no later than at the RPM/DBLM.

#### 7.3 TREATMENT COMPLIANCE

**Section 4.3 of the CTP:** Compliance will be assured by administration of all trial medication in the study centre under supervision of the investigating physician or a designee. The measured plasma concentrations will provide additional confirmation of compliance.

It is not intended to list the compliance separately. Any deviations from complete intake will be addressed in the RPM/DBLM (cf. TSAP <u>Section 6.2</u>) and described in the CTR.

#### 7.4 PRIMARY ENDPOINTS

Refer to TSAP <u>Section 7.8</u> for a description of the analysis of safety and tolerability of BI 1323495.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7.5 SECONDARY ENDPOINTS

# 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoints have been specified in the protocol.

# 7.5.2 Secondary endpoints

Section 7.3.2 of the CTP:

Assessment of dose proportionality

Dose proportionality will be assessed using the pharmacokinetic endpoints as specified in Section 5.2.2

Based on the estimate for slope parameter ( $\beta$ ), a 2-sided 90% CI for the slope will be computed. Perfect dose proportionality would correspond to a slope of 1. The assumption of a linear relationship between the log-transformed pharmacokinetic endpoint and the log-transformed dose will be checked.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

If dose proportionality over the entire dose range investigated cannot be shown, an attempt will be made to identify dose range(s), where dose proportionality can be assumed.

This analysis will be accomplished by using the XPKISTAT macro (design DB), based on the PKS.

# Graphical displays:

A regression plot will be performed, where the logarithm of dose is depicted versus logarithm of PK endpoint, including the estimated regression line from the power model and reference line of perfect proportionality ( $\beta$ =1).

TSAP for BI Trial No: 1405-0001 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report based on the TS. The date and time of drug administration will be listed for each subject.

### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

If not stated otherwise, the safety results will be sorted by treatment group.

The safety data for treated subjects who failed to complete the study (dropouts or withdrawals) will be reported as far as their data are available. All withdrawals will be documented and the reason for withdrawal recorded.

#### 7.8.1 Adverse events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature and will be based on BI standards as presented in the corporate guideline: "Analysis and Presentation of Adverse Event Data from Clinical Trials" [001-MCG-156] (2).

The standard AE analyses will be based on the number of subjects with AEs (and not on the number of AEs).

For analysis multiple AE occurrence data on the CRF will be collapsed into an AE provided that all of the following applies:

- All AE attributes are identical (lower level term (LLT), intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AE of special interest)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started within one hour after end of the first occurrence)

For further details on summarization of AE data, please refer to [001-MCG-156] (9).

#### **Section 5.2.2.1 of the CTP:** *The following are considered as AESIs:*

#### • *Hepatic injury*

A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- o an elevation of AST (aspartate aminotransferase) and/or ALT (alanine aminotransferase) ≥3-fold ULN combined with an elevation of total bilirubin ≥2-fold ULN measured in the same blood sample, or
- o aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN

These lab findings constitute a hepatic injury alert, and the subjects showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure that these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

The analysis of adverse events will be based on the concept of treatment emergent adverse events.

**Section 7.3.3 of the CTP:** The REP for BI 1323495, the time interval when measurable drug levels or PD effects are still likely to be present after administration, is not known for this first-in-human trial. Therefore, all AEs with an onset between start of treatment and the end of trial examination (last per protocol contact) will be considered on treatment.

According to ICH E3 (10), AEs classified as 'other significant' needs to be reported and will include those non-serious and non-significant adverse events with

- (i) 'action taken = discontinuation' or 'action taken = reduced', or
- (ii) marked haematological and other lab abnormalities or lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at the RPM at the latest.

An overall summary of AEs (including AESIs) will be presented.

The frequency of subjects with AEs will be summarized by treatment, primary system organ class (SOC) and preferred term (PT). Separate tables will be provided for subjects with other significant AEs according to ICH E3 (10), for subjects with serious AEs, for subjects with drug-related AEs, for subjects with drug related serious adverse events and for subjects with AESIs.

The SOC and PTs will be sorted by frequency (within SOC). The MedDRA version number will be displayed as a footnote in the respective output.

In addition, frequencies of subjects with non-serious AEs that had an incidence of > 5% for at least one treatment will be summarised by treatment, primary SOC and PT.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For disclosure of adverse events on EudraCT additional information not included in a standard AE analysis will be performed. The following three entries will be created:

- Adverse Events per arm for disclosure on EudraCT
- Non-serious Adverse Events for disclosure on EudraCT
- Serious Adverse Events for disclosure on EudraCT

### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards [001-MCG-157] (11). Tables and listings will be based on standardized values only.

Laboratory data will be analysed qualitatively via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as possible clinically significant will be flagged in the data listings.

It is the investigator's responsibility to decide whether a lab value is clinically significant abnormal or not (at the RPM/DBLM at the latest).

# 7.8.3 Vital signs

Descriptive statistics over time including change from baseline will be performed for vital signs (blood pressure and pulse rate).

#### 7.8.4 ECG

# **Continuous safety ECG monitoring (by investigator)**

Clinically relevant abnormal findings will be reported as adverse events.

No separate listing or analysis of continuous ECG monitoring will be prepared.

### 12-lead ECG

Abnormal findings will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator.

All evaluations of ECG data will be based on the TS, except the exposure-response analyses, which are based on the ECGPCS set.

### Listing of individual data

For all quantitative endpoints, listings of individual data will be shown in Appendix 16.2. For QTcB and RR only listings will be provided. Occurrences of notable findings will be flagged.

TSAP for BI Trial No: 1405-0001 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **7.8.5** Others

# Physical examination

Physical examination findings will be reported as relevant medical history/baseline condition (i.e., a condition already existent before intake of study drug) or as AE and will be summarised as such.

No separate listing or analysis of physical examination findings will be prepared.

TSAP for BI Trial No: 1405-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. **REFERENCES**

| 1. | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version. |
|---|---|
| 2. | 001-MCS-40-413: "Identify and Manage Important Protocol Deviations (iPD) ", current version, BIRDS |
| 3. | BI-KMED-COPS-TMP-0001: "iPD log", current version; KMED |
| 4. | 001-MCG-156_RD-01: "Handling of Missing and Incomplete AE Dates", current version; IDEA for CON. |
| 5. | 001-MCS-36-472_RD-01: "Noncompartmental Pharmacokinetic/Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON. |
| 6. | 001-MCG-159: "Reporting of Clinical Trials and Project Summaries", current version; IDEA for CON. |
| 7. | 001-MCS-36-472_RD-03: "Description of Analytical Transfer Files and PK/PD Data Files", current version; IDEA for CON. |
| 8. | 001-MCS 36-472: "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version; IDEA for CON. |
| 9. | 001-MCG-156: "Analysis and Presentation of Adverse Event Data from Clinical Trials", current version; IDEA for CON. |
| 10. | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version |
| 11. | 001-MCG-157: "Handling, Display and Analysis of Laboratory Data", current version; IDEA for CON. |
| 13. | BI Statistical Position Paper - Statistical Methods for PK - Reference Document 3: Regulatory recommendations for BA/BE trials and implementation instructions in clinical trial documents, version 1.0 (2017). |

TSAP for BI Trial No: 1405-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1405-0001 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1405-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1405-0001 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **HISTORY TABLE 10.**

History table Table 10: 1

| Version | Date<br>(DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Final | 10-JAN-19 | , | None | This is the final TSAP without any modification |